CLINICAL TRIAL: NCT05386186
Title: The Effect of Glimepiride Compared With Sitagliptin as an add-on Therapy to Metformin in Severe Insulin Deficiency Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University First Hospital (Other); Jiangsu Province Geriatric Institute (Unknown)
Responsible Party: Principal Investigator, Xiantong Zou, MD. Ph.D., Attending Physician of the Department of Endocrinology and Metabolism, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zhouxiantong
Record Dates: First submitted 2022-05-12; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2; Severe Insulin Deficient Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glimepiride (Experimental): All participants have background therapy of metformin 1500mg-2000mg, glimepiride1-4mg were added in the patients randomised to this arm considering the baseline HbA1c of the participants.
  Interventions: Drug: Glimepiride
- Sitagliptin (Active Comparator): All participants have background therapy of metformin 1500mg-2000mg, Sitagliptin 100mg were added in the patients randomised to this arm regardless of the baseline HbA1c level in this arm.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Glimepiride — Initiate glimepiride 1-4mg once daily as an add-on therapy to metformin and adjust the glimepiride dosage to 1-6 mg once daily in the first 12 weeks according to the diabetes management guideline recommended by the Chinese Diabetes Society.
  Other Names: SU group (sulphonylurea group)
  Arms: Glimepiride
Drug: Sitagliptin — Add sitagliptin 100mg once daily in all patients randomized to this arm.
  Other Names: DPPIVi Group (dipeptidyl peptidase IV inhibitor group)
  Arms: Sitagliptin

SUMMARY:
The purpose of the trial is to verify the effectiveness and safety of glimepiride compared with sitagliptin as an add-on therapy to metformin in severe insulin deficiency diabetes.

DETAILED DESCRIPTION:
This clinical trial is a multi-centre, prospective, intervention, randomized-controlled clinical trial, and uses a superiority test to determine whether the experimental group is superior to the control group in terms of main efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

* According to the World Health Organization (the WHO) 1999 criteria for the diagnosis of type 2 diabetes; the subtype was allocated to severe insulin deficiency diabetes (SIDD) at diagnosis using data-driven diabetes clusters APP.
* Men and women aged ≥ 18 years and ≤ 75 years;
* Diagnosed as severe insulin deficiency diabetes by the cluster classifier of Peking University People's Hospital at the initial stage of the disease course;
* Metformin monotherapy with dosage ≥1500 mg/day for at least 8 weeks;
* Diabetes duration less than 5 years;
* The HbA1c value of the central laboratory before randomization: 7.0% ≤ HbA1c <10.5%
* estimated estimated glomerular filtration rate (eGFR)>=60 ml/min1.73m2, alanine aminotransferase(ALT)<120U/L ;
* If other drugs are used during the course of the disease, these drugs should be withdrawn for more than 8 weeks;
* Without acute diabetic complications at present.

Exclusion Criteria:

* Type 1 diabetes or other special types of diabetes mellitus; glutamic acid decarboxylase antibody (GADA) positive, the subtype was allocated to other subtypes at diagnosis using data-driven diabetes clusters APP.
* Pregnancy or have a pregnancy plan within a year;
* Lactation or have a lactation plan within a year;
* Renal insufficiency, eGFR<60; transaminase elevated, ALT>= 120U/L; unstable coronary heart disease.
* Recurrent spontaneous diabetic ketosis or uncorrected acute diabetic complications;
* Participated in other clinical trials within 8 weeks before randomization; Unable to complete the study follow-up for 6 months; Have situations such as operation and need to change to insulin therapy in 6 months.
* Use concomitant medication such as glucocorticoids which can affect blood sugar.
* The investigator judged that it is not suitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of hemoglobin A1c from baseline at the end of the trial. | 26 weeks
  The Least squre mean of the decline of hemoglobin A1c from baseline to the end of the trial

SECONDARY OUTCOMES:
Hemoglobin A1c on-target rate | 26 weeks
  the percentage of A1c<7.0% or A1c<6.5%
The difference of self measure blood glucose (SMBG) at every month | for 26 weeks
  The mean of 4-point SMBG for every four weeks
The incidence rate of hypoglycemia | for 26 weeks
  Any measurement of blood glucose<3.9mmol/L or symptoms related to hypoglycemia
The level of weight gain | for 26 weeks
  The difference between body weights at the beginning and end of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Xiantong Zou, M.D. Ph.D., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Please Select, China